CLINICAL TRIAL: NCT05265988
Title: Multiparametric Assessment of Bone Response in mCRPC Patients Treated With Cabozantinib Upon Progression to Chemotherapy and Next Generation Hormonal Agents: a Phase II Study
Brief Title: Multiparametric Assessment of Bone Response in mCRPC Patients Treated With Cabozantinib
Acronym: MERIDIAN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alfredo Berruti (Other)
Responsible Party: Sponsor-Investigator, Alfredo Berruti, Director of the Medical Oncology Unit, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Organization: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASSTBS-FARM-ONC-MERIDIAN-2020
Record Dates: First submitted 2022-02-17; First posted 2022-03-04 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Carcinoma Prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabozantinib; Tablets

STUDY DESIGN:
Intervention Model Description: Monocentrici Study. The patients are treated in one arm
Masking Description: The patients are treated in one arm.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Meridian (Experimental): Cabozantinib at initial dosage of 40 mg per day and continuation of androgen deprivation therapy
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib at initial dosage of 40 mg per day and continuation of androgen deprivation therapy
  Other Names: Cabozantinib 40/20 mg tablet

SUMMARY:
Multiparametric assesment of bone response in mCRPC patients treated with Cabozantinib upon progression to chemotherapy and next generation hormonal agents: a phase II study

DETAILED DESCRIPTION:
This is a monocentric, single arm, prospective clinical trial designed to obtain explorative information about the effect of Cabozantinib on bone in prostate cancer patients with bone metastatic castration resistant disease, previously treated with two taxanes and at least one next generation hormonal agent.

Activity of bone metastatic disease will be assessed by WB-DW-MRI, while changes in bone metabolism will be studied through DXA scan and soluble biomarkers

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of prostate carcinoma,
* Age > 18 years,
* Metastatic disease documented as the presence of bone lesions o bone scan associated or not to soft tissue lesions measurable at CT/RMN,
* Eastern Cooperative Oncology Group (ECOG) performance status equal or less than 2
* Expected life expectancy ≥ 3 months,
* Patients who have already received docetaxel, cabazitaxel and at least one next generation hormonal agent (abiraterone or enzalutamide) for metastatic disease (either hormone sensitive or castration resistant),
* Subject capable to swallow the Study's medication and to comply with the Study's requirements,
* Fertile patients and their partners must agree to use methods of contraception.
* Signed informed consent.

Exclusion Criteria:

* Presence of active serious disease, active infection or co-comorbidity that may prevent the study enrollment make (at the discretion of the clinical Investigator),
* Known or suspected brain metastases or active leptomeningeal dissemination,
* History of other malignant neoplasm during the previous 5 years, different from the non-melanoma skin carcinoma,
* Absolute Neutrophil Count (ANC) < 1.500/µL, platelet < 100.000/µL, or hemoglobin < 5,6 mmol/L (< 9 g/dL) at Screening Visit (notably: patients must not receive neither any growth factor during the previous 7 days nor any blood transfusion during the 28 days preceding the hematology sampling performed at Screening),
* Total bilirubin > 1,5 x ULN at Screening Visit,
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2,5 x ULN at Screening Visit,
* Creatinine > 177 µmol/L (> 2 mg/dL) at Screening Visit,
* Albumin ≤ 30 g/L (≤ 3,0 g/dL) at Screening Visit,
* Alkaline Phosphatase ≥ 5 x ULN,
* Prothrombin time / international normalized ratio (PT/INR) or partial thromboplastin time (PTT) test ≥ 1.3 x the laboratory ULN,
* Urine protein-to-creatinine ratio (UPCR) > 1 mg/mg (or 113.0 mg/mmol) or proteinuria > 1 g/24 h,
* History of seizures or any other seizure-predisposed pathology; history of loss of consciousness or transitory ischaemic attack during the 12 months preceding the Screening visit,
* Clinically significant cardiovascular disease including:
* Myocardial infarction (6 months preceding the screening),
* Uncontrolled angina (3 months preceding the screening),
* Congestive heart failure New York Heart Association (NYHA) class 3 or 4, congestive heart failure NYHA class 3 or 4 in the past, unless a screening echocardiogram or multi-gated acquisition scan performed within three months results in a left ventricular ejection fraction that is ≥ 45%,
* History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes),
* History of long QT syndrome or corrected QT interval calculated by the Fridericia formula > 500 msec at Screening Visit,
* History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place,
* Hypotension as indicated by systolic blood pressure < 86 millimeters of mercury (mmHg) at the Screening visit,
* Bradycardia as indicated by a heart rate of < 50 beats per minute on the Screening ECG,
* Uncontrolled hypertension as indicated by systolic blood pressure > 170 mmHg or diastolic blood pressure > 105 mmHg at the Screening visit,
* History of thromboembolic events, including pulmonary embolism or untreated deep venous thrombosis (6 months preceding the screening)
* Gastrointestinal disorder affecting absorption (e.g., gastrectomy, active peptic ulcer disease within last 3 months),
* Major surgery within 8 weeks of enrollment (Day 1 Visit). Complete healing from major surgery must have occurred 4 weeks before enrollment. Complete healing from minor surgery (e.g. simple excision, tooth extraction) must have occurred at least 7 days before enrollment.
* Subjects with clinically relevant complications from prior surgery.
* Concomitant therapy with anticoagulants such as warfarin or warfarin-related agents, thrombin or coagulation factor X (FXa) inhibitors, or antiplatelet agents (e.g. clopidogrel). Low molecular weight Heparin (LMWH) and low-dose aspirin for cardioprotection (per local applicable guidelines) are permitted.
* Concomitant use of strong inhibitors of CYP3A4 (including, but not limiting to: ketoconazole, itraconazole, clarithromycin, indinavir, nefazodone, nelfinavir, and ritonavir).
* Use of herbal products that may have hormonal anti-prostate cancer activity and/or are known to decrease PSA levels (e.g., saw palmetto) or systemic corticosteroids greater than the equivalent of 10 mg of prednisone per day within 4 weeks of enrollment (Day 1 visit).
* Previously identified allergy or hypersensitivity to the study drug and/or excipients.
* Bone antiresorptive drugs (e.g., zoledronic acid or denosumab) that are started within 4 weeks of enrollment (Day 1 Visit). Bone antiresorptive drugs are permitted if already ongoing before this time point. Patients will be stratified according to zoledronic acid/denosumab exposure.
* Systemic treatment with radionuclides within 6 weeks before first dose of study treatment or radiotherapy on sites other than bone administrated within 4 weeks of enrollment (Day 1 Visit). Radiotherapy on bone administrated within 2 weeks of enrollment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible. Radiotherapy given with palliative intent will be permitted during study treatment.
* Any condition or reason that, in the opinion of the Investigator, interferes with the ability of the patient to participate in the trial, which places the patient at undue risk, or complicates the interpretation of safety data.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2024-06-29 (Actual); Study Completion 2024-06-29 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) on bone metastases through whole body diffusione weighted (WB-DW) MRI. | 6 months
  Proportion of patients attaining a partial or complete response to therapy on bone metastases by means of WB-DW MRI.

SECONDARY OUTCOMES:
Objective response rate (ORR) on bone metastases through bone scan. | 12 months.
  Proportion of patients attaining a partial or complete response to therapy on bone metastases by means of bone scan.
Quality of life through the administration of validated questionnaires. | 12 months
  Change in bone pain and quality of life through the administration of validated questionnaires.
Progression free survival (PFS). | From randomization to first evidence of progression or death from any cause.
  Time from treatment initiation and disease progression or death from any cause.
Overall survival (OS). | From randomization to death from any cause.
  Time from treatment initiation and death from any cause.
Incidence of skeletal related events (SRE). | 12 months.
  Proprtion of SRE defined as the occurrence of one among: spinal cord compression, pathologic fracture, necessity for radiation to bone or surgery to bone.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Berruti, Principal Investigator — Asst Degli Spedali Civili Di Brescia
Locations (1):
- Alfredo Berruti, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shiozawa Y, Pedersen EA, Havens AM, Jung Y, Mishra A, Joseph J, Kim JK, Patel LR, Ying C, Ziegler AM, Pienta MJ, Song J, Wang J, Loberg RD, Krebsbach PH, Pienta KJ, Taichman RS. Human prostate cancer metastases target the hematopoietic stem cell niche to establish footholds in mouse bone marrow. J Clin Invest. 2011 Apr;121(4):1298-312. doi: 10.1172/JCI43414. Epub 2011 Mar 23. PMID 21436587
- [Result] Smith M, De Bono J, Sternberg C, Le Moulec S, Oudard S, De Giorgi U, Krainer M, Bergman A, Hoelzer W, De Wit R, Bogemann M, Saad F, Cruciani G, Thiery-Vuillemin A, Feyerabend S, Miller K, Houede N, Hussain S, Lam E, Polikoff J, Stenzl A, Mainwaring P, Ramies D, Hessel C, Weitzman A, Fizazi K. Phase III Study of Cabozantinib in Previously Treated Metastatic Castration-Resistant Prostate Cancer: COMET-1. J Clin Oncol. 2016 Sep 1;34(25):3005-13. doi: 10.1200/JCO.2015.65.5597. Epub 2016 Jul 11. PMID 27400947
- [Result] Schmidt GP, Reiser MF, Baur-Melnyk A. Whole-body MRI for the staging and follow-up of patients with metastasis. Eur J Radiol. 2009 Jun;70(3):393-400. doi: 10.1016/j.ejrad.2009.03.045. Epub 2009 May 19. PMID 19457631
- [Result] Vanel D, Casadei R, Alberghini M, Razgallah M, Busacca M, Albisinni U. MR imaging of bone metastases and choice of sequence: spin echo, in-phase gradient echo, diffusion, and contrast medium. Semin Musculoskelet Radiol. 2009 Jun;13(2):97-103. doi: 10.1055/s-0029-1220880. Epub 2009 May 19. PMID 19455472
- [Result] Ma J. Dixon techniques for water and fat imaging. J Magn Reson Imaging. 2008 Sep;28(3):543-58. doi: 10.1002/jmri.21492. PMID 18777528
- [Result] Koh DM, Blackledge M, Padhani AR, Takahara T, Kwee TC, Leach MO, Collins DJ. Whole-body diffusion-weighted MRI: tips, tricks, and pitfalls. AJR Am J Roentgenol. 2012 Aug;199(2):252-62. doi: 10.2214/AJR.11.7866. PMID 22826385
- [Result] Padhani AR, Makris A, Gall P, Collins DJ, Tunariu N, de Bono JS. Therapy monitoring of skeletal metastases with whole-body diffusion MRI. J Magn Reson Imaging. 2014 May;39(5):1049-78. doi: 10.1002/jmri.24548. Epub 2014 Feb 10. PMID 24510426
- [Result] Huang W, Li X, Chen Y, Li X, Chang MC, Oborski MJ, Malyarenko DI, Muzi M, Jajamovich GH, Fedorov A, Tudorica A, Gupta SN, Laymon CM, Marro KI, Dyvorne HA, Miller JV, Barbodiak DP, Chenevert TL, Yankeelov TE, Mountz JM, Kinahan PE, Kikinis R, Taouli B, Fennessy F, Kalpathy-Cramer J. Variations of dynamic contrast-enhanced magnetic resonance imaging in evaluation of breast cancer therapy response: a multicenter data analysis challenge. Transl Oncol. 2014 Feb 1;7(1):153-66. doi: 10.1593/tlo.13838. eCollection 2014 Feb. PMID 24772219
- [Result] Senn C, Gunther B, Popp AW, Perrelet R, Hans D, Lippuner K. Comparative effects of teriparatide and ibandronate on spine bone mineral density (BMD) and microarchitecture (TBS) in postmenopausal women with osteoporosis: a 2-year open-label study. Osteoporos Int. 2014 Jul;25(7):1945-51. doi: 10.1007/s00198-014-2703-8. Epub 2014 Apr 24. PMID 24760244
- [Result] Di Gregorio S, Del Rio L, Rodriguez-Tolra J, Bonel E, Garcia M, Winzenrieth R. Comparison between different bone treatments on areal bone mineral density (aBMD) and bone microarchitectural texture as assessed by the trabecular bone score (TBS). Bone. 2015 Jun;75:138-43. doi: 10.1016/j.bone.2014.12.062. Epub 2015 Jan 6. PMID 25571842
- [Result] Shepherd JA, Schousboe JT, Broy SB, Engelke K, Leslie WD. Executive Summary of the 2015 ISCD Position Development Conference on Advanced Measures From DXA and QCT: Fracture Prediction Beyond BMD. J Clin Densitom. 2015 Jul-Sep;18(3):274-86. doi: 10.1016/j.jocd.2015.06.013. PMID 26277847
- [Result] Rosen CJ, Bouxsein ML. Mechanisms of disease: is osteoporosis the obesity of bone? Nat Clin Pract Rheumatol. 2006 Jan;2(1):35-43. doi: 10.1038/ncprheum0070. PMID 16932650
- [Result] Shapses SA, Pop LC, Wang Y. Obesity is a concern for bone health with aging. Nutr Res. 2017 Mar;39:1-13. doi: 10.1016/j.nutres.2016.12.010. Epub 2017 Jan 18. PMID 28385284
- [Result] Tang R, Ma F, Li W, Ouyang S, Liu Z, Wu J. miR-206-3p Inhibits 3T3-L1 Cell Adipogenesis via the c-Met/PI3K/Akt Pathway. Int J Mol Sci. 2017 Jul 14;18(7):1510. doi: 10.3390/ijms18071510. PMID 28708070
- [Result] Perdomo G, Martinez-Brocca MA, Bhatt BA, Brown NF, O'Doherty RM, Garcia-Ocana A. Hepatocyte growth factor is a novel stimulator of glucose uptake and metabolism in skeletal muscle cells. J Biol Chem. 2008 May 16;283(20):13700-6. doi: 10.1074/jbc.M707551200. Epub 2008 Mar 24. PMID 18362143
- [Result] Vega A, Abad S, Macias N, Aragoncillo I, Santos A, Galan I, Cedeno S, Manuel Lopez-Gomez J. Low lean tissue mass is an independent risk factor for mortality in patients with stages 4 and 5 non-dialysis chronic kidney disease. Clin Kidney J. 2017 Apr;10(2):170-175. doi: 10.1093/ckj/sfw126. Epub 2017 Feb 8. PMID 28396734
- [Result] Shepherd JA, Ng BK, Sommer MJ, Heymsfield SB. Body composition by DXA. Bone. 2017 Nov;104:101-105. doi: 10.1016/j.bone.2017.06.010. Epub 2017 Jun 16. PMID 28625918
- [Result] Martin TJ. Bone biology and anabolic therapies for bone: current status and future prospects. J Bone Metab. 2014 Feb;21(1):8-20. doi: 10.11005/jbm.2014.21.1.8. Epub 2014 Feb 28. PMID 24707463